CLINICAL TRIAL: NCT05241405
Title: Evaluation of the Impact of Taking American Ginseng for 8 Weeks on Fatigue in Patients Treated for Localized Breast or Gynecological Cancer - Randomized, Placebo-controlled, Double-blind Study
Brief Title: Evaluation of the Impact of Taking American Ginseng for 8 Weeks on Fatigue in Patients Treated for Localized Breast or Gynecological Cancer
Acronym: QISEIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: NATSUCA laboratory (Unknown); Groupement Interrégional de Recherche Clinique et d'Innovation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-A01550-41
Record Dates: First submitted 2022-02-03; First posted 2022-02-15 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer; Fatigue
Keywords: Qiseng; food supplement
MeSH Terms: conditions — Breast Neoplasms; Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Qiseng (Experimental): 200 mg/capsule of P. quinquefolius extract, i.e. 30 mg of ginsenosides, associated with 30 mg of vitamin C extracted from Camu Camu berry
  Interventions: Dietary Supplement: QISENG
- Placebo (Placebo Comparator): neutral microgranules of Qiseng® excipients without P. quinquefolius or Camu Camu extract
  Interventions: Dietary Supplement: PLACEBO

INTERVENTIONS:
Dietary Supplement: QISENG — 2 capsules/day for 8 weeks.
  Arms: Qiseng
Dietary Supplement: PLACEBO — 2 capsules/day for 8 weeks.
  Arms: Placebo

SUMMARY:
This is a multicenter randomized trial in breast cancer patients reporting cancer-related fatigue to evaluate the efficacy and safety of Qiseng® based on extract of American ginseng combined with vitamin C from extract of Camu Camu berries

ELIGIBILITY:
Inclusion Criteria:

* Patients with localized breast or gynecological cancer treated as curative adjuvant and/or neoadjuvant chemotherapy and/or adjuvant radiotherapy. These treatments must have been completed within 6 months of inclusion.

  * Patient reporting a chronic, stable fatigue state at investigator assessment, defined as a fatigue score ≥ 4 on the visual analog scale rated up to 10, experienced for at least one month
  * Maintenance therapy with hormone therapy or other maintenance therapy (trastuzumab, bevacizumab…) is allowed before and/or during the study (except for pembrolizumab, abemaciclib and PARP inhibitors, which are not authorized)
  * Patient 18 years of age or older
  * Effective contraception in women of childbearing age
  * Patient affiliated to a social security plan
  * Signed informed consent

Exclusion Criteria:

* Other identified causes of fatigue (anemia of grade > 2, underlying chronic disease known to be associated with fatigue)
* Ongoing chemotherapy (patients scheduled for oral capecitabine or trastuzumab-emtasin in the adjuvant setting are not eligible)
* Metastatic breast or gynecological cancer
* Ongoing treatment with a tyrosine kinase inhibitor or other P-gp transported molecule or Pembrolizumab or PARP inhibitors
* Patient requiring oral diabetes therapy
* Regular intake of Vitamin C (in addition to what is provided by the diet)
* Patients with chronic pain requiring daily treatment with analgesics, anti-inflammatory drugs or corticosteroids
* Consumption of ginseng-based products in the month prior to inclusion
* Hypersensitivity to any of the components of Qiseng or placebo
* Pregnant or breastfeeding patient
* Simultaneous participation in another therapeutic clinical trial (trial using an experimental product)
* Patient deprived of liberty, under guardianship or curatorship
* Patient unable to undergo the medical follow-up of the trial for geographical, social or psychopathological reasons
* History of any other malignant disease during the last 3 years, except for skin cancer other than melanoma, carcinoma in situ of the uterus. Any other solid tumor or lymphoma (without bone marrow involvement) must have been treated and show no signs of recurrence for at least 3 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2022-09-27 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Fatigue score change [min :5; max:20] | After 1 week and 4 weeks after the end of treatment (so 8 weeks of treatment)
  The difference between the initial (inclusion) score and the best score based on EORTC QLQ-FA12 questionnaire (physical fatigue dimension) between assessments at 1 week (S9) and 4 weeks (S12) after the end of treatment) will be calculated

SECONDARY OUTCOMES:
Other dimensions of fatigue [min :12; max:48] | after 4 weeks of treatment, after 8 weeks of treatment and 4 weeks after the end of treatment
  Score of emotional fatigue, cognitive fatigue, global score, according to the EORTC QLQ-FA12 self-questionnaire
The incidence of treatment-related adverse events | up to 8 weeks after the end of treatment
  The incidence of treatment-related adverse events and the number of patients in whom at least one treatment-related adverse event occurred
Quality of life level assessed by EORTC QLQ-C30 questionnaire | 4 and 8 weeks of treatment and 4 weeks after the end of treatment
  EORTC QLQ-C30 quality of life questionnaire scores
anxiety level | after 4 and 8 weeks of treatment, and 4 weeks after the end of treatment
  HADS anxiety and depression questionnaire scores
Cognitive function | after 4 and 8 weeks of treatment and 4 weeks after the end of treatment
  Cognitive function dimensions, according to the FACT-Cog self-assessment questionnaire,
Physical activity level | after 4 and 8 weeks of treatment, and again 4 weeks after the end of treatment
  measured by the IPAQ questionnaire scores
Sleep quality | after 4 and 8 weeks of treatment and 4 weeks after the end of treatment
  measured by CAT-sleep questionnaire scores
The level of acceptability of the treatment, | over a period of 8 weeks
  measured by the total number of times the treatment was taken

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - ARCOCEA_Clinique Europe, Amiens
  - Ch Bayeux, Bayeux
  - Centre Pierre Curie, Beuvry
  - Centre François Baclesse, Caen
  - Polyclinique du Parc, Caen
  - Ch Calais, Calais
  - Ch Cherbourg, Cherbourg
  - Clinique de Flandre, Coudekerque-Branche
  - Centre Henri Becquerel, Rouen
  - Clinique des Dentellières, Valenciennes

IPD SHARING:
Plan to Share IPD: No